CLINICAL TRIAL: NCT04978350
Title: Overcoming Barriers to the Uptake of Cascade Screening for Lynch Syndrome: Workbook Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of North Carolina, Chapel Hill (Other); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-3115; 1KL2TR002490-01 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-07-27 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lynch Syndrome
Keywords: Implementation Science; Cascade Screening
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Intervention Model Description: This is single arm, interventional study of 15 patients diagnosed with Lynch Syndrome and 4 genetic counselors who are working with the 15 patients.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Workbook Arm (Experimental): Participants in the Educational Workbook Arm will receive an electronic PDF version of an educational workbook via email on cascade screening in families with Lynch Syndrome. Genetic counselors will introduce the workbook to enrolled patients with Lynch Syndrome. Patient participants will use the activities and information in the workbook to communicate about Lynch Syndrome with family members.
  Interventions: Behavioral: Educational Workbook

INTERVENTIONS:
Behavioral: Educational Workbook — Let's Talk is an educational workbook on Lynch Syndrome and the benefits of cascade screening containing a series of lessons and activities on the following topics:
  What is Lynch Syndrome? Why should a patient tell a patient's family members about Lynch Syndrome? Create a list of the patient's first-degree relatives at risk for inheriting Lynch Syndrome What should a patient tell family members about Lynch Syndrome? Create a script for the patient to use in discussing Lynch Syndrome with family What are common concerns the patient might hear from family members? How should the patient tell family members about Lynch Syndrome? Create a plan and goals for the patient to reach out to family members What the patient should do if conversation with family is difficult What are common terms and questions about Lynch Syndrome? How can the patient manage having Lynch Syndrome? Where can the patient find additional information about living with Lynch Syndrome?

SUMMARY:
The investigators will evaluate the feasibility of an intervention to improve Lynch syndrome cascade screening uptake. The investigators will conduct a pilot study among 15 patients diagnosed with Lynch Syndrome and 5 genetic counselors to assess the feasibility and intermediate outcomes of an educational workbook containing exercises and resources to improve family communication among individuals with Lynch Syndrome and first-degree relatives of individuals with Lynch Syndrome.

DETAILED DESCRIPTION:
Genetic counselors of patients with Lynch Syndrome and patients with Lynch Syndrome will test a planning tool (referred to as an educational workbook) for cascade screening. Five genetic counselors and 15 patients with Lynch Syndrome will be recruited from the UNC Health System and the Ohio State Comprehensive Cancer Center. Genetic counselors will identify patients with Lynch Syndrome and introduce the study opportunity to potential patient participants. All patients and genetic counselors will complete a telephone enrollment call and provide informed consent to participate. Enrolled patients will work with enrolled genetic counselors to complete the first workbook exercise and then patients will complete the remaining exercises alone for over approximately 1 month. After genetic counselors and patients have completed using the workbook, the investigators will conduct qualitative virtual interviews over Zoom and a post-intervention electronic survey to understand the participants' experiences using the workbook. The investigators aim to understand the feasibility of using the workbook as an intervention in clinical practice to improve genetic testing uptake in families with Lynch Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with Lynch Syndrome within the last 365 days.
* Patients and genetic counselors must be age 18 or older.
* Patients must be receiving care from genetic counselors at Ohio State University Comprehensive Cancer Center or at UNC Health System.
* Genetic counselors must provide Lynch Syndrome counseling for patient participants at Ohio State University Comprehensive Cancer Center or at UNC Health System.
* Patients and genetic counselors must be able to speak and read in English.
* Patients and genetic counselors must review informed consent documents and provide verbal consent to participate in the study.

Exclusion Criteria: There are no exclusion criteria for study participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Roberts, PhD, Principal Investigator — UNC Eshelman School of Pharmacy
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 08/01/2021 through 04/02/2024 at one cancer center in North Carolina.
Pre-assignment Details: A total of 20 subjects consented and started to the study.
Groups:
- Educational Workbook Arm: Participants will receive an electronic PDF version of an educational workbook via email on cascade screening in families with Lynch Syndrome.
Period: Overall Study
Arm/Group | Educational Workbook Arm
Started | 20
Completed | 14
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: The participants consented and started the study activities.
Arm/Group | Educational Workbook Arm
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  <18 years old | 0
  18-40 years old | 5
  41- 64 years old | 10
  Unknown | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
  Unknown/Not reported | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Workbook Assessed Through Likert Score Scale
Description: Participants evaluated the workbook using seven acceptability criteria rated on a 5-point Likert scale, where 1 indicated "Strongly Disagree" and 5 indicated "Strongly Agree." The criteria assessed ease of use, clarity of exercises, enjoyment, usefulness for understanding Lynch Syndrome, support for communicating genetic information, time acceptability, and overall satisfaction. Each participant's responses were summed up to produce a total acceptability score ranging from 7 to 35, with higher scores indicating greater acceptability. A score of 28 or higher (80% of the maximum score, which was 35) was defined as an acceptable intervention.
Time Frame: Post 4 Weeks of Workbook Use
Population: Participants who joined the study and responded to the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Workbook Arm
Number analyzed (Participants) | 13
Participants
  score is higher the threshold | 10
  score is below the threshold | 3

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
Arm/Group | Educational Workbook Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT04978350/Prot_SAP_001.pdf